CLINICAL TRIAL: NCT06421610
Title: Implementation and Evaluation of Pressurized Intrathoracic Aerosol Chemotherapy (PITAC) for the Treatment of Patients With Malignant Pleural Effusion. A Danish Phase I Study (OPC5 Study)
Brief Title: OPC5: Pressurized IntraThoracic Aerosol Chemotherapy (PITAC) in Patients With Malignant Pleural Effusion.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PITAC-OPC5
Record Dates: First submitted 2023-04-26; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Malignant Pleural Effusion; Pleural Neoplasms; Quality of Life; Chemotherapy Effect; Chemotherapeutic Toxicity; Pleural Carcinomatosis; Pleural Cavity Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Neoplasms; Pleural Effusion

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PITAC (Experimental): Malignant Pleural Effusion (MPE) from colorectal or appendix cancer will be treated with Pressurized IntraThoracic Aerosol Chemotherapy (PITAC) using oxaliplatin 92 mg/m2 in 150 ml dextrose. MPE from non-colorectal or -appendix cancer will be treated with PITAC using cisplatin 10.5 mg/m2 in 150 ml saline and 2.1 mg/m2 in 50 ml saline.
  PITAC is performed with a intrapleural pressure of 12 mmHg and the aerosolised chemotherapy will be nebulized at a maximum pressure of 300 PSI and a flow-rate of 0.5-1.8 ml/min. The PITAC directed treatment will be planned with 4 week intervals and patients may receive bi-directional systemic chemotherapy simultaneously.
  Interventions: Drug: PITAC

INTERVENTIONS:
Drug: PITAC — Cisplatin, oxaliplatin and doxorubicin are standard, commercially available intravenous cytostatic drugs in oncologic treatment with alkylating and topoisomerase inhibitor effect, respectively. Based on the available data and experience from 11 PITAC procedures at OPC, PITAC with cisplatin, oxaliplatin and doxorubicin for intrapleural administration is expected to be well tolerated with a minimal of nausea, subcutaneous emphysema and transient chest pains.

SUMMARY:
This study will monitor and evaluate patient and personnel safety and toxicity during the implementation and evaluation of Pressurized IntraThoracic Aerosol Chemotherapy (PITAC) directed treatment. Furthermore, this study will focus on Quality of Life questionnaires, LENT score, and evaluate pain and breathlessness using af visual analogue scales (VAS).

DETAILED DESCRIPTION:
This is a safety and feasibility study of repeated (minimum two procedures) PITAC directed treatments, and the primary outcome is the number of patients with medical adverse events (AEs) according to the Common Terminology Criteria for Adverse Events (CTCAE) and/or surgical complications according to the Clavien-Dindo classification. This study will include consecutive MPE patients until 20 patients have completed at least two PITAC´s. The PITAC directed treatment will be performed in 4 week intervals. Bedside ultrasound, VAS-pain and VAS-breathlessness, and Quality of Life questionnaires will be performed at baseline, one month follow-up and three months follow-up.

Patients with MPE who are eligible for surgery are identified during the multidisciplinary tumor (MDT) conference at the Department of Surgery, Odense University Hospital (OUH), and included based on predefined in- and exclusion criteria. Patients with MPE from non-colorectal or -appendix cancer will be treated with a combination of cisplatin and doxorubicin. Patients with MPE from colorectal or appendix cancer will be treated with oxaliplatin.

In brief, The PITAC procedure is the application of aerosolized chemotherapy into the pleural cavity using thoracoscopy. PITAC is performed in the prone or lateral position. A double lumen endotracheal tube is used to allow exclusion of the ipsilateral lung, but this is not (always) necessary with the patient in the prone position. The first trocar is placed guided by ultrasound, and after safe positioning a second trocar can be inserted guided by video thoracoscopy. The chemotherapy is applied to the pleural cavity through a nebulizer inserted through one of the trocars and linked to a high-pressure injector. After five minutes the chemotherapy has been delivered to the pleural cavity, and after an additional 30 minutes of simple diffusion, the intrathoracic air saturated with chemotherapy is evacuated through a series of filters.

The patients are monitored for a minimum of one day and will after each PITAC directed treatment be screened for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic MPE visible with bedside ultrasound
* Histologically or cytologically verified malignancy
* Status CT-scan not older than four weeks
* MPE requiring at least one drainage procedure
* Drained ≥ 14 days before the first PITAC directed treatment
* Bidirectional systemic chemotherapy or immunotherapy ≥ 14 days before the first PITAC directed treatment or no simultaneous systemic chemotherapy or immunotherapy
* ECOG Performance status 0-2
* Life expectancy ≥ 3 months
* Age ≥ 18 years
* Danish-speaking and reading patients
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* A history of allergic reaction to cisplatin or other platinum containing compounds or doxorubicin
* Renal impairment, defined as GFR < 40 ml/min (Cockcroft-Gault Equation)
* Myocardial insufficiency, defined as NYHA class > 2
* Impaired liver function defined as bilirubin ≥1.5
* Fertility, pregnancy and lactation: Female subjects will be considered of non-reproductive potential if they are either a, b or c:

  1. postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age a high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
  2. have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 6 weeks prior to screening.
  3. have a congenital or acquired condition that prevents childbearing. Previous intrathoracic chemotherapy, intrathoracic antibody treatment or chemical pleurodesis
* Any other condition or therapy, which in the investigator´s opinion may pose a risk to the patient or interfere with the study objects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Medical adverse events | 30 days from PITAC directed treatment
  Number of patients with medical adverse events (AEs) according to the Common Terminology Criteria for Adverse Events (CTCAE) version 6.0 defined as CTCAE ≥ 4 within 30 days after the procedure.
Surgical complications | 30 days from PITAC directed treatment
  Number of patients with surgical complications according to the Clavien-Dindo classification defined as Clavien-Dindo ≥ 3b within 30 days after the procedure.

SECONDARY OUTCOMES:
Number of patients completing three PITAC treatments | 12 months
  To evaluate the number of patients completing three PITAC treatments
Extent of visible pleural metastasis | 12 months
  To macroscopically evaluate the extent of visible pleural metastasis (PLM) during PITAC directed therapy via the new PLM-score based on size of lesions (LS).
  LS 0 No tumor seen LS1 Tumor up to 0.5 cm LS2 Tumor up to 5.0 cm LS3 Tumor > 5.0 cm or confluence
Pathology on pleural metastasis biopsies | 12 months
  To evaluate Pleural Regression Grade Score (Ple-RGS) in biopsies from visible pleural metastasis Ple-RGS is a modification of the Peritoneal Regression Grading score (PRGS). Ple-RGS 1: Complete histological response Ple-RGS 2: Regressive changes are predominant over cancer cells (major response) Ple-RGS 3: Cancer cells are predominant over regressive changes (minor response) Ple-RGS 4: No response
Cytology on malignant pleural effusion fluid | 12 months
  To evaluate cytology on MPE during PITAC directed therapy. The cells will be graded according to a five-tiered score: malignant cells, suspicious cells, atypical cells, no malignant cells and other
LENT score | 12 months
  To evaluate the LENT score after each PITAC directed therapy. Low risk: 0-1 Moderate risk: 2-4 High risk: 5-7
Length of Stay (LOS) | 12 months
  Quantify the length of stay (LOS) (surgery = day 0)
Personnel safety (environmental) | 12 months
  Assess personnel safety by measuring of platinum traces in the operating room.
Personnel safety (biological) | 12 months
  Assess personnel safety by measuring of platinum traces in blood samples from surgeons and/or OR nurses.
Lung function evaluation by SAT | 12 months
  To evaluate lung function by saturation (SAT) before PITAC directed treatment (day 0) and at discharge (day 1), day 30 and 3 months after the last PITAC directed treatment
Breathlessness | 12 months
  To evaluate breathlessness using visual analogue scales (VAS-breath) before PITAC directed treatment (day 0) and at discharge (day 1), day 30, and 3 months after the last PITAC directed treatment
Pain assessment | 12 months
  To evaluate pain using visual analogue scales (VAS-pain) before PITAC directed treatment (day 0) and at discharge (day 1), day 30, and 3 months after the last PITAC directed treatment
Quality of Life questionnaires | 12 months
  To evaluate the quality of life with EORTC-QLQ-C30 at baseline, day 30 and 3 months after the last PITAC directed treatment
Change in MPE volume | 12 months
  To calculate the change in volume of drained MPE from 2 months before the first PITAC treatment to three months after the last PITAC treatment
Long term complications | 12 months
  To assess long-term complications 3 months after the third PITAC directed treatment
Survival | 12 months
  Median overall survival
Lung function evaluation by FEV1 | 12 months
  To evaluate lung function by Forced Expired Volume in the first second (FEV1) before PITAC directed treatment (day 0) and at discharge (day 1), day 30 and 3 months after the last PITAC directed treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Odense PIPAC Center, Department of Surgery, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
Publications and presentations will be based on patient data, but the database is not open to other researchers.